CLINICAL TRIAL: NCT06811142
Title: EVALUATION OF THE EFFECTS OF EARLY APPLICATION OF BOTULINUM TOXIN IN PATIENTS WITH A FIRST CEREBRAL VASCULAR EVENT.
Brief Title: Early Botulinum Toxin for Muscle Stiffness Reduction in First-Time Stroke Patients: Improving Recovery and Independence
Acronym: EARLY BOT-SPAS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Roberto Carlos Pech Arguelles, principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-3201-072
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Spasticity; Stroke; Neurological Rehabilitation
Keywords: NEUROPLASTICITY; Post-Stroke Spasticity; Stroke Rehabilitation; Early Intervention; Botulinum Toxin (BoNT-A); Modified Ashworth Scale
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; abobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: This study uses a Parallel Assignment Model with two groups: an intervention group receiving early botulinum toxin (BoNT-A) injections and a control group undergoing standard rehabilitation without the toxin. The intervention aims to prevent spasticity-related complications by leveraging early treatment during the neuroplastic phase, within 12 weeks post-stroke. Randomized and controlled conditions will ensure unbiased results, with outcomes measured over short, medium, and long-term follow-up periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- intervention (Active Comparator): Participants in the intervention group will receive early botulinum toxin type A (BoNT-A) injections in addition to a standard rehabilitation program. The botulinum toxin will be administered within the first 12 weeks following stroke onset, targeting muscles affected by spasticity. The injections aim to reduce abnormal muscle tone, prevent contractures, and improve functional mobility. Rehabilitation therapy will include physical exercises, range-of-motion activities, and muscle-strengthening interventions tailored to individual recovery needs. The combined therapy is designed to optimize motor function, promote neuroplasticity, and improve overall independence and quality of life.
  Interventions: Drug: Botulinum Toxin Type A (BoNT-A)
- control (No Intervention): Participants in the control group will undergo a standard rehabilitation program without the early application of botulinum toxin. The rehabilitation will consist of physical therapy focused on improving muscle strength, range of motion, and functional independence. Treatment will be tailored to each participant's condition and recovery progress, following established post-stroke rehabilitation protocols. This group will serve as the comparator to evaluate the additional benefits of early botulinum toxin intervention.

INTERVENTIONS:
Drug: Botulinum Toxin Type A (BoNT-A) — This intervention involves the early administration of botulinum toxin type A (BoNT-A) within the first 12 weeks after a cerebrovascular event. The injections target muscles affected by spasticity, aiming to reduce abnormal tone, prevent contractures, and improve functional mobility. BoNT-A works by blocking acetylcholine release at the neuromuscular junction, resulting in muscle relaxation. Ultrasound guidance or anatomical landmarks will be used for accurate injection. This early intervention capitalizes on the neuroplastic window and is combined with standard rehabilitation to enhance motor recovery and prevent long-term complications.
  Other Names: Botulinum Neurotoxin A; BoNT-A; AbobotulinumtoxinA
  Arms: intervention

SUMMARY:
This study examines the early use of botulinum toxin in patients recovering from their first stroke to help reduce muscle stiffness and improve mobility. Spasticity, a condition that causes abnormal muscle tightness, is a common complication following strokes. It can result in decreased independence, pain, joint contractures, and difficulty performing daily activities. Early intervention is critical to prevent long-term complications and improve recovery outcomes.The participants are men and women aged 18 and older who have recently experienced their first stroke. These patients, admitted to the Regional General Hospital No. 1 "Lic. Ignacio García Téllez" in Mérida, Yucatán, will receive botulinum toxin injections alongside a comprehensive rehabilitation program. Botulinum toxin, commonly known for its muscle-relaxing effects, will be administered within the first three months after the stroke. This early timeline aims to maximize recovery by addressing muscle tightness before it worsens.The study will evaluate how the combination of botulinum toxin and physical therapy affects muscle tone, functional independence, and overall quality of life. Key measurements include the Modified Ashworth Scale (MAS) to assess muscle stiffness, the Barthel Index to evaluate daily activity independence, and cognitive assessments to monitor brain recovery. Patients' progress will be tracked over several months to measure the intervention's short, medium, and long-term impact.Previous research suggests that early application of botulinum toxin can prevent long-lasting muscle contractures and improve mobility, but more studies are needed to confirm its benefits in stroke rehabilitation. The results of this research could help establish early botulinum toxin injections as a standard practice in stroke recovery programs, reducing disability and healthcare costs while improving the lives of stroke survivors.

DETAILED DESCRIPTION:
This clinical study evaluates the impact of early application of botulinum toxin on patients experiencing their first cerebrovascular event. Spasticity, characterized by abnormal muscle stiffness and involuntary muscle contractions, is a frequent complication of strokes that can lead to reduced mobility, pain, joint deformities, and a diminished ability to perform daily activities. The study aims to determine whether early intervention with botulinum toxin, in combination with rehabilitation therapy, can mitigate the development and severity of post-stroke spasticity, improve muscle tone, and enhance functional outcomes.

Patients eligible for participation include men and women aged 18 and older, admitted with a confirmed diagnosis of a recent stroke within the first seven days of symptom onset. The intervention will involve botulinum toxin injections administered within the early subacute phase (up to 12 weeks post-stroke) to maximize the neuroplastic window and reduce the risk of permanent muscle contractures. The study will be conducted over three years at the Regional General Hospital No. 1 "Lic. Ignacio García Téllez," Mérida, Yucatán.

The primary outcomes assessed will include changes in muscle tone, evaluated by the Modified Ashworth Scale (MAS), and functional independence, measured using the Barthel Index. Secondary outcomes will assess quality of life, cognitive performance, and overall rehabilitation progress through tools such as the Mini-Mental State Examination (MMSE) and the Fugl-Meyer Assessment Scale. The study design is a prospective, controlled clinical trial comparing patients receiving early botulinum toxin injections with those undergoing standard rehabilitation only.

This research aims to provide valuable clinical evidence regarding the effectiveness of early botulinum toxin application in preventing long-term disabilities, enhancing recovery, and reducing healthcare burdens associated with post-stroke spasticity. By identifying clinical predictors of spasticity, the study will contribute to the development of targeted, time-sensitive interventions that optimize stroke rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years old. Beneficiaries treated in the Emergency and/or Internal Medicine service at HGR No. 1, IMSS Mérida, Yucatán, with an acute stroke confirmed by clinical symptoms and a new ischemic lesion detected through magnetic resonance imaging or computed tomography within 7 days of onset.

Exclusion Criteria:

* Severe cognitive deficits.

  * Severe language comprehension disorders.
  * Lack of capacity to give informed consent.
  * Physical disability already existing before the acute stroke.
  * Subarachnoid hemorrhage.
  * Transient ischemic attack.
  * Any other neurological disorder that could affect muscle tone (Conditions related to the spine, brain infection and traumatic brain injury).
  * Any amputation of the limb on the affected side.
  * Peripheral neuropathy of the upper and/or lower limbs.
  * Patients who have suffered a previous stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Baseline (within 7 days post-stroke) 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The Modified Ashworth Scale (MAS) is a 6-point ordinal scale (0, 1, 1+, 2, 3, 4) used to assess spasticity by evaluating resistance during passive movement of a joint. The scoring system is as follows:
  0: No increase in muscle tone.
  1: Slight increase in tone, with a catch and release or minimal resistance at the end of the range of motion.
  1+: Slight increase in tone, with a catch followed by minimal resistance throughout less than half of the range of motion.
  2: More marked increase in tone through most of the range, but the joint moves easily.
  3: Considerable increase in tone, making passive movement difficult. 4: Affected part is rigid in flexion or extension.
MODIFIED TARDIEU SCALE | Baseline (within 7 days post-stroke) 8 weeks post-intervention 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The Modified Tardieu Scale (MTS) assesses spasticity by measuring muscle response to passive stretching at different velocities. It evaluates both the angle of muscle reaction (R1) and the final range of motion (R2). The key feature of the MTS is its sensitivity to velocity-dependent resistance, distinguishing it from the Modified Ashworth Scale. Joint movement is tested at three speeds: slow (V1), normal (V2), and fast (V3). The difference between R1 and R2 reflects dynamic spasticity and muscle stiffness.
  The scale assigns qualitative scores (0-5) based on the severity of the muscle reaction:
  0: No resistance throughout the movement.
  1. Slight resistance with no clear catch.
  2. Clear catch at a precise angle, followed by release.
  3. Fatigable clonus with fewer than 10 seconds of contraction.
  4. Unfatigable clonus lasting more than 10 seconds.
  5. Joint is immobile.

SECONDARY OUTCOMES:
MINI MENTAL STATE EXAMINATION | Baseline (within 7 days post-stroke) 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The Mini-Mental State Examination (MMSE) is a widely used screening tool to assess cognitive function, often employed in stroke rehabilitation studies to monitor neurological recovery. The test evaluates five cognitive domains: orientation, immediate memory, attention and calculation, recall, and language. It includes tasks such as recalling objects, following commands, and answering orientation questions. The MMSE is scored out of 30 points, with higher scores indicating better cognitive function.
  A score of 24 or higher is generally considered normal, while scores below this threshold suggest varying degrees of cognitive impairment. The MMSE will be administered at different intervals to assess how early intervention with botulinum toxin and rehabilitation affects patients' cognitive recovery. Its role as a secondary outcome helps determine whether improvements in motor function correlate with cognitive benefits during stroke rehabilitation.
BARTHEL INDEX | Baseline (within 7 days post-stroke) 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The Barthel Index is a standardized tool used to assess a patient's level of independence in performing basic activities of daily living (ADLs). It evaluates 10 tasks, including feeding, bathing, dressing, using the toilet, walking, and controlling bladder and bowel movements. Each task is scored based on the patient's ability to perform the activity independently or with assistance. The total score ranges from 0 to 100, with higher scores indicating greater independence.
  0 points: Complete dependence 100 points: Full independence
NIHSS SCALE | BASELINE 1 month post-intervention
  The NIHSS Scale is a clinical tool used to assess the severity of neurological deficits in patients who have experienced a stroke. It evaluates multiple domains, including level of consciousness, motor function, sensory abilities, language, coordination, and visual fields. The scale consists of 15 items, each scored from 0 to 4, with a maximum score of 42 indicating severe stroke and a score of 0 indicating no neurological deficits.
  Key categories assessed include:
  Motor Function: Arm and leg movement Sensory Function: Response to tactile stimuli Language and Speech: Aphasia or dysarthria Level of Consciousness: Alertness and responsiveness
Modified Rankin Scale | Baseline (within 7 days post-stroke) 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The Modified Rankin Scale (mRS) is a 7-point ordinal scale used to measure functional status and the degree of disability or dependence in activities of daily living following a stroke. It evaluates outcomes ranging from no symptoms (0) to severe disability or death (6). The scale is widely used in stroke rehabilitation to monitor recovery and assess long-term functional outcomes.
  Scoring:
  0: No symptoms.
  1. No significant disability; able to carry out all usual activities.
  2. Slight disability; unable to perform all previous activities but manages without assistance.
  3. Moderate disability; requires some help but can walk without assistance.
  4. Moderately severe disability; unable to walk or attend to bodily needs without assistance.
  5. Severe disability; requires constant nursing care and attention.
  6. Death.
Fugl-Meyer Upper and Lower Extremity Scale | Baseline (within 7 days post-stroke) 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The Fugl-Meyer Assessment (FMA) for Upper and Lower Extremities is a widely used, validated tool to evaluate motor recovery after stroke. It assesses motor function, balance, sensation, and joint movement through a series of tasks designed to measure impairments in the affected limbs. The assessment is divided into two parts:
  1. Upper Extremity (FMA-UE) Focuses on shoulder, elbow, wrist, hand, and coordination tasks. Tasks are scored from 0 (no function) to 2 (normal function) based on movement ability, precision, and control.
     Maximum score: 66 points for the upper limb.
  2. Lower Extremity (FMA-LE) Evaluates hip, knee, and ankle movement, including weight-bearing tasks and reflex activity.
  Similar scoring from 0 to 2 per task, with a maximum score of 34 points for the lower limb.
  Key Areas Assessed:
  Voluntary Movement: Flexion, extension, and joint movement. Coordination and Speed: Smoothness and accuracy of movements.
Goal Attainment Scaling | Baseline (within 7 days post-stroke) 6 months post-intervention 12 months post-intervention
  Goal Attainment Scaling (GAS) is an individualized, patient-centered tool used to measure the extent to which a patient achieves predetermined rehabilitation goals. It involves setting specific, measurable goals tailored to the patient's condition, which can include improvements in motor function, independence, pain reduction, or daily activities. Each goal is rated on a 5-point scale, ranging from -2 to +2, where:
  * 2: Much less than expected outcome.
  * 1: Somewhat less than expected outcome. 0: Expected outcome achieved.
    * 1: Somewhat better than expected outcome.
    * 2: Much better than expected outcome.
MEDICAL RESEARCH COUNCIL | Baseline (within 7 days post-stroke) 12 weeks post-intervention 6 months post-intervention 12 months post-intervention
  The MRC Scale is a validated clinical tool used to assess muscle strength in patients with neurological or muscular impairments, such as after a stroke. It evaluates the ability of specific muscle groups to generate force against resistance. Each muscle group is tested, and strength is graded on a 6-point ordinal scale (0 to 5):
  0: No muscle contraction observed.
  1. Flicker of contraction, but no visible joint movement.
  2. Active movement possible only with gravity eliminated.
  3. Active movement against gravity, but no resistance.
  4. Active movement against gravity and some resistance.
  5. Normal strength, full movement against maximum resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Regional No.1 "Lic. Ignacio García Téllez" IMSS, Calle 41 101, Fénix, 97155 Mérida, Yuc., Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kong KH, Lee J, Chua KS. Occurrence and temporal evolution of upper limb spasticity in stroke patients admitted to a rehabilitation unit. Arch Phys Med Rehabil. 2012 Jan;93(1):143-8. doi: 10.1016/j.apmr.2011.06.027. PMID 22200394
- [Result] Opheim A, Danielsson A, Alt Murphy M, Persson HC, Sunnerhagen KS. Early prediction of long-term upper limb spasticity after stroke: part of the SALGOT study. Neurology. 2015 Sep 8;85(10):873-80. doi: 10.1212/WNL.0000000000001908. Epub 2015 Aug 14. PMID 26276377
- [Result] Sunnerhagen KS. Predictors of Spasticity After Stroke. Curr Phys Med Rehabil Rep. 2016;4:182-185. doi: 10.1007/s40141-016-0128-3. Epub 2016 Jul 22. PMID 27547509
- [Result] Zeng H, Chen J, Guo Y, Tan S. Prevalence and Risk Factors for Spasticity After Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2021 Jan 20;11:616097. doi: 10.3389/fneur.2020.616097. eCollection 2020. PMID 33551975
- [Result] Rosales RL, Efendy F, Teleg ES, Delos Santos MM, Rosales MC, Ostrea M, Tanglao MJ, Ng AR. Botulinum toxin as early intervention for spasticity after stroke or non-progressive brain lesion: A meta-analysis. J Neurol Sci. 2016 Dec 15;371:6-14. doi: 10.1016/j.jns.2016.10.005. Epub 2016 Oct 11. PMID 27871449
- [Result] Patel AT, Ward AB, Geis C, Jost WH, Liu C, Dimitrova R. Impact of early intervention with onabotulinumtoxinA treatment in adult patients with post-stroke lower limb spasticity: results from the double-blind, placebo-controlled, phase 3 REFLEX study. J Neural Transm (Vienna). 2020 Dec;127(12):1619-1629. doi: 10.1007/s00702-020-02251-6. Epub 2020 Oct 27. PMID 33106968
- [Result] 11. Stephen, AD (sf). Spasticity in adults: management using botulinum toxin. Royal College of Physicians, 3-22.
- [Result] Francisco GE, Balbert A, Bavikatte G, Bensmail D, Carda S, Deltombe T, Draulans N, Escaldi S, Gross R, Jacinto J, Ketchum N, Molteni F, Moraleda S, ODell MW, Reebye R, Satero P, Verduzco-Gutierrez M, Walker H, Wissel J. A practical guide to optimizing the benefits of post-stroke spasticity interventions with botulinum toxin A: An international group consensus. J Rehabil Med. 2021 Jan 1;53(1):jrm00134. doi: 10.2340/16501977-2753. PMID 33057730
- [Result] Sunnerhagen KS, Opheim A, Alt Murphy M. Onset, time course and prediction of spasticity after stroke or traumatic brain injury. Ann Phys Rehabil Med. 2019 Nov;62(6):431-434. doi: 10.1016/j.rehab.2018.04.004. Epub 2018 May 16. PMID 29753889
- [Result] Ganguly J, Kulshreshtha D, Almotiri M, Jog M. Muscle Tone Physiology and Abnormalities. Toxins (Basel). 2021 Apr 16;13(4):282. doi: 10.3390/toxins13040282. PMID 33923397
- [Result] Li S, Francisco GE, Rymer WZ. A New Definition of Poststroke Spasticity and the Interference of Spasticity With Motor Recovery From Acute to Chronic Stages. Neurorehabil Neural Repair. 2021 Jul;35(7):601-610. doi: 10.1177/15459683211011214. Epub 2021 May 12. PMID 33978513
- [Result] Glaess-Leistner S, Ri SJ, Audebert HJ, Wissel J. Early clinical predictors of post stroke spasticity. Top Stroke Rehabil. 2021 Oct;28(7):508-518. doi: 10.1080/10749357.2020.1843845. Epub 2020 Nov 6. PMID 33156735
- [Result] 4. Marlenne, RS (2015). In-hospital mortality due to cerebrovascular diseases in the main public health institutions in Mexico. CONAMED-PAHO BULLETIN, 7-11
- [Result] 3. Cuadrado, A. (2009). Stroke rehabilitation: assessment, prognosis and treatment. Galicia Clinic/Galician Society of Internal Medicine, 25-34.
- [Result] Cantu-Brito C, Majersik JJ, Sanchez BN, Ruano A, Quinones G, Arzola J, Morgenstern LB. Hospitalized stroke surveillance in the community of Durango, Mexico: the brain attack surveillance in Durango study. Stroke. 2010 May;41(5):878-84. doi: 10.1161/STROKEAHA.109.577726. Epub 2010 Apr 1. PMID 20360543
- [Result] 1. Parra, JA (2019). Ischemic stroke: extensive review of the literature for the primary care physician. Med Int Méx, 61-63.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT06811142/Prot_SAP_ICF_000.pdf